CLINICAL TRIAL: NCT00397111
Title: Development of Functional and Structural Magnetic Resonance Imaging Techniques for the Study of Mood and Anxiety Disorders
Brief Title: Development of Magnetic Resonance Imaging Techniques for Studying Mood and Anxiety Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070021; 07-M-0021
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-25

CONDITIONS: Mood Disorders; Anxiety Disorders
Keywords: Morphometry; BOLD; fMRI; Spectrometry; Relaxometry; Natural History; Healthy Volunteer; HV
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer: Healthy Volunteer/control group
  Interventions: Device: 7T Magnetic Resonance Imaging scanner
- Major Depressive Disorder: Individuals with Major Depressive Disorder
  Interventions: Device: 7T Magnetic Resonance Imaging scanner

INTERVENTIONS:
Device: 7T Magnetic Resonance Imaging scanner — Non-significant risk device used for brain imaging

SUMMARY:
This study is intended to help develop new MRI imaging techniques for studying mood and anxiety disorders. Researchers believe that depression and anxiety disorders may cause structural and functional changes in the brain. This study will optimize the way MRI scans are collected to look at brain structure and examine how the brain behaves while subjects perform particular tasks. Healthy volunteers and individuals with major depressive disorder may be eligible for this study.

Participants undergo magnetic resonance imaging (MRI) and neuropsychological testing. : Individuals will be asked to participate in an MRI study on one of several scanners. The scanner used will measure blood flow in the brain, concentrations of certain chemicals in the brain, or magnetic properties of the brain. The scan may involve They watching a screen presenting images or doing a task in which they respond to pictures or sounds. Participants may be asked to return for additional scans.

The study also involves neuropsychological tests, which assess cognitive performance. Often, people with mood disorders have subtle changes in performance on these tests that allow researchers to pinpoint where brain abnormalities occur. Before the tests can be used in patients, they must be validated by using healthy subjects. These tests are presented either orally, in written form, or on a computer.

DETAILED DESCRIPTION:
Objective

A major component of understanding the pathogenesis of mood and anxiety disorders is expected to involve elucidation of abnormalities in brain structure and function associated with these conditions. Historically post-mortem histopathological and neurochemical assessments constituted the primary methods for investigating abnormalities of brain structure and function in psychiatric disorders. However, the significance of the results from such studies has been limited by the relatively poor availability of specimens from subjects with mood and anxiety disorders who had been unmedicated and clinically well-characterized antemortem. By allowing for in vivo human studies, medical imaging technologies provide efficient, accurate, and non-invasive alternatives for characterizing brain structure and function. The recent rapid development of magnetic resonance imaging (MRI) technology, in particular, has provided powerful tools for assessing a wide range of cerebral physiological and morphological characteristics. To optimally exploit the potential of these rapidly evolving MRI scanning and hardware capabilities in investigations of mood and anxiety disorders, new techniques and applications must be developed and tested. The technical development protocol proposed herein will assess new imaging techniques and hardware, and will develop novel cognitive tasks for application in the study of mood and anxiety disorders. The primary objective of this protocol is the development of MRI experiments for characterizing the physiological correlates of mood and anxiety disorders. In addition, the pilot projects encompassed within this protocol involve the optimization of existing MRI pulse sequences, the application of new pulse sequences for structural and functional MR imaging, and the development of new functional MRI (fMRI) tasks that can elucidate neural function within the cognitive-behavioral domains affected in mood and anxiety disorders. This protocol will also allow testing of existing imaging hardware that can increase the spatial resolution, contrast, and sensitivity of MR images. Such hardware includes the use of multi-channel radio frequency (RF) coils and patient monitoring equipment. Development of these techniques and applications will directly enhance the sensitivity and specificity of MRI studies of mood and anxiety disorders.

Study Population

This study will involve 250 healthy volunteers and 90 patients with major depressive disorder.

Design

This technical development protocol will assess new imaging techniques and hardware, and will develop novel cognitive tasks for application in the study of mood and anxiety disorders. Subjects will have the option to participate in one or several procedures conducted under this protocol, including fMRI, Magnetic Resonance Spectroscopy (MRS), Magnetoencephalography (MEG), behavioral tasks, and rating scales.

Outcome Measures

Primary outcome measures on neuropsychological tests will include parameters such as accuracy and reaction time. Secondary outcome measures will include differences in reaction time or accuracy between different testing conditions. Outcome measures from MRI scanning sessions will include signal-to-noise ratio, contrast-to-noise ratio, structural volumes, metabolite concentrations (in the case of MRS), relaxation times (in the case of relaxometry), and BOLD time series (in the case of fMRI).

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Controls

* Male and female subjects between 18 and 65 years of age
* Subjects must be able to give written informed consent prior to participation in this study.
* Subjects who do not currently meet and have never met criteria for any major psychiatric disorder, and who have no known first degree relatives with mood disorders.
* For cognitive experiments utilizing language stimuli only native English speakers will be enrolled.

Major Depressive Disorder

* Male and female subjects between 18 and 65 years of age.
* Subjects have been found eligible for other ETPB research protocols according to 01-M-0254.
* Subjects must fulfill DSM-IV or V criteria for Major Depression based on clinical assessment and confirmed by a structured diagnostic interview (SCID-P).
* Subjects must be able to give written informed consent prior to participation in this study.
* For cognitive experiments utilizing language stimuli, only native English speakers will be enrolled.

EXCLUSION CRITERIA:

Healthy Control

* Subjects with major medical or neurological disorders expected to influence cerebral blood flow or morphology, or taking any medication that is likely to influence the imaging parameters-of-interest within 3 weeks of scanning.
* Women who are pregnant are excluded from the study. Subjects will undergo pregnancy testing no more than 24 hours prior to MRI scanning.
* Subjects with contraindication to MRI scanning such as aneurysm clips, implanted neural stimulator, implanted cardiac pacemaker or auto-defibrillator, cochlear implant, or ocular foreign body.
* A history of drug or alcohol abuse within 1 year or a lifetime history of drug or alcohol dependence (DSM-IV) or alcohol use disorder (DSM-V equivalent).

Major Depressive Disorder

* Presence of Axis 1 psychiatric diagnosis other than Major Depression or an Axis 2 disorder
* Subjects with major medical or neurological disorders expected to influence cognitive function or are taking any drugs likely to affect mood or cognitive function within 1 week of study participation. Depressed subjects will not be tapered/withdrawn from medications under this study.
* A history of drug or alcohol abuse within 1 year or a lifetime history of drug or alcohol dependence (DSM-IV) or alcohol use disorder (DSM-V equivalent).
* Subjects with major medical or neurological disorders expected to influence cerebral blood flow or morphology.
* Women who are pregnant or breastfeeding will be excluded from MRI portions of the study. Subjects will undergo pregnancy testing no more than 24 hours prior to MRI scanning.
* Subjects with contraindication to MRI scanning such as aneurysm clips, implanted neural stimulator, implanted cardiac pacemaker or auto-defibrillator, cochlear implant, or ocular foreign body.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult healthy volunteers and individuals with major depressive disorder will be recruited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2006-12-06 (Actual)

PRIMARY OUTCOMES:
BOLD time series | Varies based on experiment
  Magnetic Resonance Imaging data
Structural volumes | Varies based on experiment
  Magnetic Resonance Imaging data
Accuracy | Varies based on experiment
  Neuropsychological testing data
Contrast-to-noise ratio | Varies based on experiment
  Magnetic Resonance Imaging data
Signal-to-noise ratio | Varies based on experiment
  Magnetic Resonance Imaging data
Relaxation times | Varies based on experiment
  Reflexometry data
Metabolite concentrations | Varies based on experiment
  Magnetoencephalography data
Reaction time | Varies based on experiment
  Neuropsychological testing data

SECONDARY OUTCOMES:
Reaction time between testing conditions | Varies based on experiment
  Neuropsychological testing data
Accuracy between testing conditions | Varies based on experiment
  Neuropsychological testing data

CONTACTS AND LOCATIONS:
Overall Officials: Allison C Nugent, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical, demographic, and phenotype participant data collected during the trial, after deidentification.
Supporting Information: SAP, Analytic Code
Time Frame: Sharing my start at any time during data collection, no later 1 year following completion of the study.
Access Criteria: Fully de-identified data may be shared on publicly available data repositories. The PI will review additional requests for data not shared in repositories.

REFERENCES:
- [Background] Drevets WC, Price JL, Simpson JR Jr, Todd RD, Reich T, Vannier M, Raichle ME. Subgenual prefrontal cortex abnormalities in mood disorders. Nature. 1997 Apr 24;386(6627):824-7. doi: 10.1038/386824a0. PMID 9126739
- [Background] Drevets WC, Ongur D, Price JL. Neuroimaging abnormalities in the subgenual prefrontal cortex: implications for the pathophysiology of familial mood disorders. Mol Psychiatry. 1998 May;3(3):220-6, 190-1. doi: 10.1038/sj.mp.4000370. PMID 9672897
- [Background] Drevets WC. Neuroimaging and neuropathological studies of depression: implications for the cognitive-emotional features of mood disorders. Curr Opin Neurobiol. 2001 Apr;11(2):240-9. doi: 10.1016/s0959-4388(00)00203-8. PMID 11301246
- [Derived] Lamontagne SJ, Gilbert JR, Zabala PK, Waldman LR, Zarate CA Jr, Ballard ED. Clinical, behavioral, and electrophysiological profiles along a continuum of suicide risk: evidence from an implicit association task. Psychol Med. 2024 May;54(7):1431-1440. doi: 10.1017/S0033291723003331. Epub 2023 Nov 24. PMID 37997749
- [Derived] Lally N, An L, Banerjee D, Niciu MJ, Luckenbaugh DA, Richards EM, Roiser JP, Shen J, Zarate CA Jr, Nugent AC. Reliability of 7T (1) H-MRS measured human prefrontal cortex glutamate, glutamine, and glutathione signals using an adapted echo time optimized PRESS sequence: A between- and within-sessions investigation. J Magn Reson Imaging. 2016 Jan;43(1):88-98. doi: 10.1002/jmri.24970. Epub 2015 Jun 7. PMID 26059603
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2007-M-0021.html